CLINICAL TRIAL: NCT05882799
Title: Ultrasound-guided vs. Blinded Dry Needling for Piriformis Syndrome: A Randomized Trial
Brief Title: Ultrasound-guided vs. Blinded Dry Needling for Piriformis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Priformis1
Record Dates: First submitted 2023-05-07; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided dry needling group (Active Comparator): Patients in this group will receive dry needling for piriformis syndrome under real-time ultrasound guidance.
  Interventions: Procedure: Ultrasound-guided dry needling
- Blinded dry needling group (Active Comparator): Patients in this group will receive dry needling for piriformis syndrome without ultrasound guidance.
  Interventions: Procedure: Blinded dry needling

INTERVENTIONS:
Procedure: Ultrasound-guided dry needling — Ultrasound-guided dry needling is a minimally invasive technique that involves inserting a sterile acupuncture needle into trigger points of a muscle while monitoring the needle's progress with real-time ultrasound imaging. In this technique, a trained practitioner visualizes the piriformis muscle and the surrounding structures using an ultrasound machine, and then inserts the needle through the skin and into the muscle tissue, guided by the ultrasound image.
  Arms: Ultrasound-guided dry needling group
Procedure: Blinded dry needling — Blinded dry needling is a minimally invasive technique that involves inserting a sterile acupuncture needle into trigger points of a muscle without using real-time imaging guidance. In this technique, the practitioner relies solely on their palpation skills to locate the trigger points of the piriformis muscle and inserts the needle through the skin and into the muscle tissue.
  Arms: Blinded dry needling group

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of ultrasound-guided versus blinded dry needling for the treatment of piriformis syndrome.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the efficacy of ultrasound-guided versus blinded dry needling for the treatment of piriformis syndrome. Patients in both groups will receive three weekly sessions of dry needling performed by a single experienced physiatrist. The intervention will involve inserting a sterile acupuncture needle into the trigger points of the piriformis muscle and manipulating the needle to elicit a twitch response. Patients in the ultrasound-guided group will receive dry needling under real-time ultrasound guidance, while patients in the blinded group will receive dry needling without ultrasound guidance. Patients will be assessed before treatment, after treatment, after the third week, and after three months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-65 years.
* Clinical diagnosis of piriformis syndrome based on the following criteria: buttock pain, radiating pain to the posterior thigh, and tenderness over the piriformis muscle.
* Pain intensity of at least 4 out of 10 on a visual analog scale (VAS).
* Willingness to comply with the study protocol and provide informed consent.

Exclusion Criteria:

* Previous surgery or injection therapy for piriformis syndrome.
* Contraindications to dry needling, such as bleeding disorders or skin infections.
* Pregnancy or breastfeeding.
* History of neurological disorders, such as sciatica, radiculopathy, or neuropathy.
* History of serious psychiatric illness or substance abuse.
* Inability to complete the study questionnaires or follow-up assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale for Pain | First day, after three weeks, after three months
  A Visual Analog Scale (VAS) for pain is a commonly used tool to measure the intensity of pain experienced by a patient. It typically consists of a horizontal or vertical line, typically 10 centimeters long, with endpoints labeled as "no pain" and "worst possible pain." The patient is asked to mark on the line the point that best represents the intensity of their pain, with the distance from the "no pain" end of the line to the patient's mark representing the pain score.
Change in Oswestry Disability Index (ODI) | First day, after three weeks, after three months
  The Oswestry Disability Index (ODI) is a self-administered questionnaire that is widely used to assess the functional status of patients with low back pain or sciatica. The ODI consists of 10 sections, each relating to a different aspect of functional impairment, such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. Each section is scored on a scale of 0-5, with a total score ranging from 0 (no disability) to 50 (complete disability). The ODI is a validated and reliable tool for assessing functional status and has been used in many clinical trials to evaluate the effectiveness of interventions for low back pain or sciatica.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon reasonable request by the corresponding author.
Supporting Information: Study Protocol, CSR
Time Frame: 1 month.
Access Criteria: Individual participant data will be shared upon reasonable request by the corresponding author.